CLINICAL TRIAL: NCT04491331
Title: Hemodynamic Changes Due to Prone Position in Healthy Volunteers
Brief Title: Hemodynamic Changes Due to Prone Position
Status: Completed | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, Principal investigator, University Hospital Hradec Kralove
Other Study IDs: UH HradecKralove
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Hemodynamics Instability; Prone Position
Keywords: hemodynamics; prone position; cardiac output
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-anesthetized volunteers: Hemodynamic parameters will be measured in supine position. Volunteers will be turned into prone position. After a five-minute stabilization phase will be monitored CI, MAP, heart rate (HR), stroke volume variation SVV, systemic vascular resistance index (SVRI) by non-invasive measurements using a ClearSight (Edwards) in two prone positions (lying on support system allowing a free abdomen and then lying flat without any device). Furthermore, the width of the inferior vena cava and vena jugularis interna, vena saphena and vena cephalica will be measured by ultrasound. The measurement will be performed in inspiration and in expiration phase.
  Interventions: Procedure: prone position

INTERVENTIONS:
Procedure: prone position — Unsupported prone position with arms along the body in neutral position will be used first without any supportive device except support of heels with a soft cylindrical device, head will be held in a neutral position using prone head rest. After recording of all measered values, the prone position using the prone position support system will be tested. The support system allows free movement of the lower thorax and abdomenal wall, upper arms are elevated and angled in 90 degrees (in shoulders and elbows). Heels will be positioned at the level of the heart using a supportive cylindrical device. Head will be held in a neutral position using prone head rest.

SUMMARY:
Perioperative prone position may be associated with hemodynamic instability. The causes of instability have not yet been precisely elucidated. The aim of this study is to demonstrate physiological changes during prone positioning in healthy volunteers .

DETAILED DESCRIPTION:
The prone position could decrease the cardiac index (CI), mainly due to reduction in stroke volume, with little changes in heart rate. Mean arterial pressure (MAP) could be maintained by increased systemic vascular resistance (SVR) in the majority of patients.

The aim of this study is to describe hemodynamic changes in two different surgical prone positions in 10 healthy non-anesthetized volunteers (flat position and using a support system allowing a free abdomen) by non-invasive measurement of hemodynamics (ClearSight, Edwards) and indirectly evaluated intra-abdominal pressure using ultrasound. The ClearSight system provides advanced hemodynamic parameters (cardiac index CI, stroke volume SV, stroke volume variation SVV, systemic vascular resistance SVR, mean arterial pressure MAP) from a finger cuff.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years,
* American Society of Anesthesiologists (ASA) Physical Status Classification I
* agreement with study participation

Exclusion Criteria:

* disagreement with study participation,
* BMI over 40
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 6 male and 6 female healthy, non-anesthetized volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Cardiac Index | 5 minutes
  after changing supine to prone position

SECONDARY OUTCOMES:
Changes in vena cava diameter | 5 minutes
  after changing supine to prone position
Changes in vena jugularis diameter | 5 minutes
  after changing supine to prone position
Changes in vena saphena diameter | 5 minutes
  after changing supine to prone position
Changes in vena cephalica diameter | 5 minutes
  after changing supine to prone position

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Kukralova, MD, Study Director — UH Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kukrálová L, Dostálová V, Dostál P. Hemodynamic changes in prone position - a non-invasive physiological study. Anest. intenziv. Med.. 2021;32(2):82-86. doi: 10.36290/aim.2021.010.